CLINICAL TRIAL: NCT02363790
Title: Primary Fascial Closure With Laparoscopic Ventral Hernia Repair: A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Mike K Liang, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-14-0170
Record Dates: First submitted 2015-02-02; First posted 2015-02-16 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Hernia, Ventral
Keywords: Ventral Hernia; Laparoscopic
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bridging LVHR (Other): Laparoscopic ventral hernia repair without closure of central defect (bridging repair)
  Upon completion of the lysis of adhesions, the margins of the hernia defect will be measured and marked. The hernia defect size will be measured with the abdomen completely desufflated and insufflated at 15 mm Hg externally (on the skin).
  A coated mesh with at least four cm of overlap on all sides will be placed. Mesh will be secured with at least four but no more than eight trans-fascial sutures. Titanium tacks will be placed in a double crown technique where tacks are placed every 1 cm on the periphery and every 3 cm along the fascial edge (bridged or closed).
  Interventions: Procedure: Bridging LVHR
- LVHR PFC (Other): Ventral hernia repairs in the primary fascial group will be performed similarly except prior to placement of the mesh, the defect will be closed. After the defect size is measured, the mesh will be chosen based upon the unclosed defect size and size will not be adjusted. The hernia defect will be closed as described previously 9,10 with 0-prolene transfascial sutures placed every 1-2 cm. The two caudal-most and cranial-most sutures will be placed. The abdomen will be desufflated and these sutures will be secured. The abdomen will be reinsufflated to 15 mm Hg and the defect progressively closed. Upon completion of fascial closure, the mesh will be placed in the standard fashion as describe above. The lateral overlap will be increased due to the fascial closure.
  Interventions: Procedure: LVHR PFC

INTERVENTIONS:
Procedure: LVHR PFC — Information included in arm description
  Other Names: Trancutaneous closure of the central defect
  Arms: LVHR PFC
Procedure: Bridging LVHR — Information included in arm description
  Other Names: standard LVHR
  Arms: Bridging LVHR

SUMMARY:
This study is comparing the outcomes patients undergoing LVHR, PFC as opposed to a bridged repair with assessment of patient reported satisfaction and function at 6 months of follow-up.

DETAILED DESCRIPTION:
Introduction: While randomized controlled trials have demonstrated that laparoscopic ventral hernia repair (LVHR) as compared to open repair is associated with decreased rates of surgical site infection (SSI) and shorter lengths of hospital stay, the adoption of LVHR has been limited. Less than one-fourth of ventral hernias are repaired with a laparoscopic approach in the United States. One of the main reasons cited for the lack of widespread adoption of LVHR is failure to improve patient symptoms. Following LVHR, up to 70% of patients continue to complain of an abdominal bulge and one-third of patients complain of poor function. The investigators have previously reported that primary fascial closure (PFC) with LVHR is feasible and when compared to case-matched controls, PFC improved outcomes of recurrence, bulging, and patient function.

Hypotheses: Primary Hypothesis: In patients undergoing LVHR, PFC as opposed to a bridged repair will improve patient reported satisfaction and function at 1 year of follow-up. Secondary Hypotheses: (1) PFC is safe and feasible to perform by general surgeons facile at LVHR. Compared to bridged LVHR, (2) PFC will decrease recurrence rates and (3) PFC will decrease the rate of clinician-diagnosed eventration following LVHR.

Methods: A randomized controlled trial to compare the outcomes of two methods of LVHR: bridged repair with mesh or PFC with mesh will be performed. PFC is estimated to improve patient satisfaction and patient function from composite scores on the validated and hernia-specific Modified Activities Assessment Scale (best score of 100). We expect the change in score (1 year mAAS score minus baseline scores) of the two groups to be 40 and 26 with a standard deviation of 25. Assuming a two-sided alpha of 0.05 and beta of 0.20, and 20% dropout rate, 120 patients will need to be randomized (n=60/group). The investigators' healthcare system performed 300 LVHRs last year. The investigators anticipate being able to accrue the sample size in 12 months.

Randomization and Allocation: In the operating room, prior to mesh placement, the patient will be randomized using a computer-generated sequence in variable permuted blocks. Allocation will be through a phone call to the study office. We chose to stratify the patient by hernia defect size instead of stratifying by baseline PCO.

Data Collection and Outcomes: A surgeon blinded to the treatment allocation will perform post-operative assessment at 14 days, 30 days, and 1 year post-operative. The primary outcome of change in patient-reported satisfaction and function will be assessed through the validated, hernia-specific survey, modified Activities Assessment Scale. Secondary outcomes will include all intra-operative complications related to PFC, hernia recurrence, clinician-assessed eventration, and any Dindo-Clavien 2-5 complication. Other patient reported outcomes assessed include likelihood to undergo the surgery again, likelihood to recommend surgery to their family or friends, and levels of pain.

Analysis: The primary outcome will be compared using Wilcoxon Rank Sum test. A Bayesian analysis will be performed to determine the posterior point estimates, credible intervals, and probability to decrease hernia recurrence with PFC will be calculated. In order to refine the study, when half of the expected patients (88) completed 1 year follow up we performed a blinded interim power analysis. We compared the change in PCO between the two groups and refined the sample size. Based upon these findings, the sample size was decreased from 176 to 120 patients.

Anticipated Results: This study will provide patients and providers with high-quality information on the risks and benefits of PFC versus bridging repair in LVHR. If efficacious, a multi-center effectiveness trial to assess long-term outcomes such as hernia recurrence can be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Patient desires an elective surgical repair,
2. patient is able to give informed consent,
3. diagnosis of a midline ventral hernia with a fascial defect width on clinical examination or CT scan of 3-10 cm in size,
4. body mass index <40kg/m2,
5. candidate for LVHR based upon surgeon assessment.

Exclusion Criteria:

1. acute or urgent presentation,
2. multiple defects defined as defects from two separate incisions,
3. patient has loss of domain assessed,
4. patient has a severe co-morbid condition likely to limit survival to <2 years,
5. contamination noted pre-operative or intra-operative,
6. patient is pregnant or intends to become pregnant during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction and function | 12 months
  Change in patient satisfaction and function evaluated through the modified Activities Assessment Scale, a validated, hernia-specific score that can be compared pre- and post-operative

SECONDARY OUTCOMES:
Surgical site infection | 30 days after surgery
  Surgical site infection will be defined by the Center for Disease Control and Prevention (CDC) definition of a surgical site infection.
Hernia recurrence and clinical bulging/eventration | 2 years after surgery
  number of patients with a clinical hernia recurrence: A clinician blinded to the treatment allocation will determine if the patient has a clinical hernia recurrence defined as any palpable defect of the anterior abdominal wall.
  -Radiographic hernia recurrence: If the clinical team orders a CT scan, results of a radiographic hernia recurrence will be reported. Radiographic hernia recurrence will be defined as any defect of the anterior abdominal wall and will be determined by a blinded radiologist and surgeon not part of the clinical care team.
Clinical bulging/eventration | 2 years after surgery
  number patients with clinical bulging/eventration: Clinician reported eventration: A study coordinator blinded to the treatment allocation will determine if the patient has clinical eventration defined as any bulge of tissue or mesh beyond the natural contour of the abdomen on supine flexion.
  -Patient reported eventration: A study coordinator blinded to the treatment allocation will ask the patient if they feel that they still have their hernia bulge.

CONTACTS AND LOCATIONS:
Overall Officials: Mike K Liang, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (5):
- United States (5):
  - George Washington University, Washington D.C., District of Columbia
  - University of Iowa, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - University of Nevada at Las Vegas, Las Vegas, Nevada
  - Lyndon B. Johnson General Hospital, Houston, Texas

REFERENCES:
- [Derived] Bernardi K, Olavarria OA, Holihan JL, Kao LS, Ko TC, Roth JS, Tsuda S, Vaziri K, Liang MK. Primary Fascial Closure During Laparoscopic Ventral Hernia Repair Improves Patient Quality of Life: A Multicenter, Blinded Randomized Controlled Trial. Ann Surg. 2020 Mar;271(3):434-439. doi: 10.1097/SLA.0000000000003505. PMID 31365365